CLINICAL TRIAL: NCT05641701
Title: Stimulation of the Thalamus to Ameliorate Persistent Disfluency: Pilot Study
Brief Title: Stimulation of the Thalamus to Ameliorate Persistent Disfluency
Acronym: SToPeD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Professor of Neurosurgery, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-02984
Record Dates: First submitted 2022-11-23; First posted 2022-12-08 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Persistent Developmental Stutter; Childhood-Onset Fluency Disorder (Stuttering)
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Childhood-Onset Fluency Disorder; Stuttering

STUDY DESIGN:
Intervention Model Description: Each participant will act as their own control. Each individual's stutter will be assessed with DBS system OFF (control) and DBS ON (treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Simulation (DBS) System (Experimental): The DBS device will be turned on to compare stutter to when the device was off (which would be the control).
  Interventions: Device: System On; Device: System off

INTERVENTIONS:
Device: System On — The DBS system will be turned on, and the individual's stutter will be assessed.
Device: System off — The DBS system will be turned off, and the individual's stutter will be assessed.

SUMMARY:
Persistent developmental stutter / childhood onset fluency disorder is a disabling condition leading to significant communication and psychological disability. Established treatment consists of intensive speech therapy, and whilst initially effective, has a waning long-term benefit.

Our research team aims to provide evidence of stutter management by addressing the primary neurological issue in this disorder using Deep Brain Stimulation. The investigators propose to perform bilateral DBS on 3 participants with stutter refractory to intensive speech therapy, to determine a response in their stutter. The assessments will be double-blinded. The investigators will use the outcome of this small pilot study to determine the feasibility and details of a larger randomized controlled trial.

DETAILED DESCRIPTION:
Suitable participants are referred by speech pathology centers, after having failed an intensive speech therapy program. Referred participants are contacted by the Neurosurgery DBS Clinic, and assessed for suitability and willingness to participate.

These potential participants will be contacted by the DBS Clinic at Vancouver General Hospital to discuss the scope of the study, and educate them about deep brain stimulation. Those who wish to be included in the study will attend a face-to-face appointment at the DBS Clinic.

At the initial appointment, informed consent will take place. Baseline assessments will be undertaken, including the Overall Assessment of the Speaker's Experience of Stuttering (OASES), Voice-related Quality of Life (VRQoL), and "The One Page Stuttering Assessment". The participants will be referred for a functional MRI for mapping of speech and language laterality.

The participants will then undergo surgery for implantation of a bilateral thalamic DBS system. They will stay overnight in the hospital, and have a post-operative CT scan on the first post-operative day. This scan will be used to assess accuracy of electrode placement, as per usual technique.

4 weeks post-operatively, the participants will attend the DBS Clinic for programming of their devices.

4 weeks after device programming, the participants will attend the DBS clinic for 1-page stutter assessment with bilateral electrodes on, bilateral electrodes off, left electrode on, and right electrode on, as well as OASES and VRQoL.

The scores from the 1-page stutter assessment, as well as pre- and post-operative OASES and VRQoL, will be compared via the Wilcoxan rank sum test for nonparametric repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 19 and 76 years old
* Individuals with persistent developmental stutter refractory to intensive speech therapy, as diagnosed by a speech and language therapist.

Exclusion Criteria:

* Children and adolescents will not be included, as there is a significant percentage of developmental stuttering that will spontaneously resolve in this age group.
* Patients who have not trialed standard therapy will not be included in this study.
* Patients with mild symptoms.
* Patients who have a neurodegenerative disease.
* Patients with a bleeding diathesis.
* Patients who are unable to communicate.

MRI Specific Exclusion criteria:

* Patients with a cardiac pacemaker or defibrillator.
* Patient with an insulin or infusion pump.
* Patients with a cochlear, otologic, or ear implant.
* Patients with an implant held in place by a magnet.
* Patients with tissue expanders.
* Patients with implanted clips, catheters, clamps, valves, or other metal.
* Patients with tattoos or permanent makeup above shoulders.
* Patients with shrapnel or other retained metal.
* Patients who are pregnant.

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Change of One-Page Suttering Assessment from Baseline to Post-Operation | Baseline assessment will be done pre-operatively. Four weeks after device programming, the patients will attend the DBS clinic for 1-page stutter assessment with bilateral electrodes on.
  Objectively assesses individual's stutter. Divide the number of instances of stuttering by the number of syllables in the sample and multiply by 100 to obtain the percentage of stuttered syllables.

SECONDARY OUTCOMES:
Change of Voice Related Quality of Life (VRQoL) from Baseline to Post-Operation | Baseline assessment will be done pre-operatively. Four weeks after device programming, the patients will attend the DBS clinic with bilateral electrodes on to asses quality of life post surgery.
  A 10-question, 5 point rating scale assessment, with higher scores reflecting a worse subjective voice-related quality of life.
Change of Overall Assessment of the Speaker's Experience of Stuttering (OASES) from Baseline to Post-Operation | Baseline assessment will be done pre-operatively. Four weeks after device programming, the patients will attend the DBS clinic with bilateral electrodes on to asses subjective voice experience post surgery.
  5-point scale that indicates the amount of adverse impact a person experiences due to stuttering, with higher scores indicating higher levels of negative impact.